CLINICAL TRIAL: NCT03787875
Title: Impact of Periodontal Treatment on the RANKL/OPG Ratio in Crevicular Fluid
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Andres Lopez Roldan, Associate professor, University of Valencia
Other Study IDs: UV2
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Periodontal Diseases; Biomarkers; Bone Resorption
Keywords: RANKL; OPG; periodontal biomarkers; alveolar bone loss; chronic periodontitis
MeSH Terms: conditions — Periodontal Diseases; Bone Resorption; Alveolar Bone Loss; Chronic Periodontitis | interventions — Periodontal Index

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: The control group included 10 periodontally healthy subjects without signs or symptoms of periodontal disease.
- Study: The study group included 15 subjects diagnosed with mild or advanced chronic periodontitis. Each periodontal patient had one non-affected single-rooted tooth (healthy site) and another single-rooted tooth with periodontitis (periodontitis site) with the following features:
  Healthy site: a single-rooted tooth with probing depths below or equal to 3 mm without recession and without bleeding on probing.
  Periodontitis site: another single-rooted tooth from the same patient with clinical attachment loss equal to or greater than 6 mm and bleeding upon probing.
  Interventions: Procedure: periodontal treatment

INTERVENTIONS:
Procedure: periodontal treatment — In the study group, periodontal scaling and root planning treatment of the 4 quadrants was performed for two consecutive weeks without the use of antiseptics or antibiotics, and the patients were instructed in oral hygiene, including both brushing techniques and proximal hygiene.
  Groups: Study

SUMMARY:
Objectives: Alveolar resorption is one of the most important events in periodontitis. Osteoclast activity is regulated by the ratio between receptor activator of NF-κB ligand (RANKL) and osteoprotegerin (OPG). The aim of this study was to evaluate changes in the RANKL/OPG ratio in crevicular fluid after periodontal treatment.

Material and methods: A total of 15 patients with periodontitis were included in the study group. Samples were collected from an area with active periodontitis and a healthy area. The RANKL and OPG levels were measured before and after periodontal scaling and root planing (SRP) treatment. The study group was compared to the control group, which included 10 patients without periodontitis.

DETAILED DESCRIPTION:
Material and methods Study design A case-control study was proposed. A group of periodontally healthy subjects was compared to a group of patients with periodontitis before and after scaling and root planing.

Two sites were studied in each subject with periodontitis: one affected site (with periodontitis) and one healthy site (without periodontal disease); the latter site served as a control. Thus, the study units were the healthy and pathological sites before and after SRP treatment.

The masking was triple blind, including the researcher in charge of sample collection, the laboratory technician and the statistician.

Due to the absence of pre-established reference values for the RANKL and OPG concentrations in periodontal health, the results obtained were compared to a control group of subjects with periodontally healthy conditions during the second part of the study.

This protocol was approved by the ethics committee of the University of Valencia (Spain) according to the Declaration of Helsinki. Written informed consent was obtained from the study subjects.

Sample selection The sample size was determined in relation to the main variable (the RANKL and OPG concentrations); currently, no reference values are available for the concentrations of these parameters under healthy or periodontal disease conditions. Therefore, to determine the sample size, the investigators used the results of previously published studies. Bostanci et al. (2011) and Buduneli et al. (2009) (sample sizes of 27 and 20 subjects, respectively) analysed the concentration changes of these parameters in the CVF before and after basic periodontal treatment.

Therefore, 25 subjects were included in the final sample in our study. The subjects were recruited consecutively at the Periodontics Unit at the Faculty of Medicine and Odontology of the University of Valencia.

The control group included 10 periodontally healthy subjects without signs or symptoms of periodontal disease.

The study group included 15 subjects diagnosed with mild or advanced chronic periodontitis. Each periodontal patient had one non-affected single-rooted tooth (healthy site) and another single-rooted tooth with periodontitis (periodontitis site) with the following features:

Healthy site: a single-rooted tooth with probing depths below or equal to 3 mm without recession and without bleeding on probing.

Periodontitis site: another single-rooted tooth from the same patient with clinical attachment loss equal to or greater than 6 mm and bleeding upon probing.

The exclusion criteria were as follows: subjects with aggressive periodontitis; systemic diseases or consumption of drugs affecting bone metabolism; antibiotic, anti-inflammatory or contraceptive treatment for the last three months prior to study initiation; antiplatelet therapy for the last 7 days prior to study onset; primary or secondary occlusal trauma; periapical or periodontal abscess in some of the teeth included in the study; any type of periodontal treatment within the last 6 months; under orthodontic treatment; smoking; and pregnant or breastfeeding.

Periodontal clinical examination:

The examination was performed by only one explorer using a Williams type manual periodontal probe (PQ-OW 208 396, Hu-Friedy®, USA). The probing depth, recession and attachment loss were measured for six sites per tooth. The "Gingival Bleeding Index" of the six sites per tooth was used to assess bleeding upon probing. The Silness and Loe index was used to assess dental plaques.

A complete radiographic series (18 radiographs) was performed for the study group with the ORing paralleling system (Dentsply®) and digital phosphor plates (Durr dental ®). Two bitewing horizontal radiographs were taken in the control group.

Periodontal treatment In the study group, periodontal scaling and root planning treatment of the 4 quadrants was performed for two consecutive weeks without the use of antiseptics or antibiotics, and the patients were instructed in oral hygiene, including both brushing techniques and proximal hygiene. Four weeks after the last SRP, the patients were examined clinically, and samples of crevicular fluid were collected again.

Study sequence Day 0- Subjects were chosen based on the inclusion and exclusion criteria. Crevicular fluid samples were collected.

Day 7- CVF samples were collected from the selected sites in both groups, and the samples were processed.

Day 14- Periodontal treatment (study group): scaling and root planing of 2 quadrants and provision of oral hygiene instructions.

Day 21- Periodontal treatment (study group): scaling and root planing of the 2 remaining quadrants and provision of oral hygiene instructions.

Day 49- Control group: clinical record and crevicular fluid sample collection and processing.

Collection of crevicular fluid The Periotron® 8000 was calibrated prior to sample collection [27]. In the study group, 4 CVF samples were collected, 2 for each single-rooted tooth with the clinical conditions described above. Two samples from one single-rooted tooth were collected from the control group.

Supragingival plaque was removed with a sterile curette, sluiced, isolated with cotton rolls and dried with air to avoid contamination with saliva. The tip of the Periopaper® was inserted into the sulcus or periodontal pocket until resistance was found and maintained for 30 seconds; tips dyed with blood were discarded. Subsequently, the CVF volume was measured by the Periotron 8000®.

In the following step, each sample was allocated into a sterilised Eppendorf tube with 100 microlitres of buffer containing phosphate-buffered saline (PBS) with protease inhibitors (C.N. P8340 Sigma, MO, USA). The Eppendorf tubes were centrifuged at 15,000 rpm for 5 min; then, another 100 microlitres of buffer was added, and the tubes were centrifuged for 5 min at 15,000 rpm. Finally, 200 microlitres of each sample was stored at -80°C prior to processing.

Sample processing RANKL and OPG were quantified using an enzyme-linked immunosorbent assay (ELISA). The technical specifications of the RANKL (total Human ELISA, BioVendor) and OPG (Bender MedSystems) kits were followed. The total RANKL and OPG concentrations were assessed.

ELIGIBILITY:
Inclusion Criteria:

1. -The control group included:

   * 10 periodontally healthy subjects
   * Without signs or symptoms of periodontal disease.
2. -The study group included:

   * 15 subjects diagnosed with mild or advanced chronic periodontitis.
   * One non-affected single-rooted tooth (healthy site)
   * Single-rooted tooth with periodontitis (periodontitis site) with the following features: with clinical attachment loss equal to or greater than 6 mm and bleeding upon probing.

Exclusion Criteria:

* Subjects with aggressive periodontitis
* Systemic diseases or consumption of drugs affecting bone metabolism
* Antibiotic, anti-inflammatory or contraceptive treatment for the last three months prior to study initiation
* Antiplatelet therapy for the last 7 days prior to study onset
* Primary or secondary occlusal trauma
* Periapical or periodontal abscess in some of the teeth included in the study
* Periodontal treatment within the last 6 months
* Orthodontic treatment
* Smoking
* Pregnant or breastfeeding.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is the classic refreshing race of the population of Spain.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2016-06-05 (Actual); Study Completion 2016-11-06 (Actual)

PRIMARY OUTCOMES:
Levels of RANKL in crevicular fluid | 49 days
  receptor activator of NF-κB ligand.RANKL is a protein that determines the activation of osteoclasts by binding to the RANK membrane receptor that preosteoclates possess.
  The ranks wi be measured in μg / μl.
Levels of OPG in crevicular fluid | 49 days
  osteoprotegerin.Osteoprogesterian is a soluble protein that acts as a decoy blocked RANK receptor and thus initiating osteoclastogenesis.
  The opg will be measured in μg / μl.

SECONDARY OUTCOMES:
probing depth | 49 days
  Probing depth, is the distance from the free gingival margin to the bottom of the periodontal pocket. This parameter will be measured in mm.
clinical attachment level | 49 days
  Is the distance from the free cementoenamel junction to the bottom of the periodontal pocket. This parameter will be measured in mm.
bleeding upon probing | 49 days
  Percentage of points with bleeding on probing in relation to the total number of points probed.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez Roldan A, Garcia Gimenez JL, Alpiste Illueca F. Impact of periodontal treatment on the RANKL/OPG ratio in crevicular fluid. PLoS One. 2020 Jan 27;15(1):e0227757. doi: 10.1371/journal.pone.0227757. eCollection 2020. PMID 31986169